CLINICAL TRIAL: NCT02203019
Title: PRO-DEFENSE: Propofol Versus Dexmedetomidine for Sedation in Mechanically Ventilated Patients With Sepsis
Brief Title: Study of Sedative Medications in Patients With Severe Infection and Respiratory Failure
Acronym: PRO-DEFENSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L14-136
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Sepsis; Respiratory Failure; Agitation
Keywords: Dexmedetomidine; Propofol; Sepsis; Mechanical Ventilation; Respiratory Failure
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency; Psychomotor Agitation | interventions — Propofol; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): Propofol will be administered for sedation.
  Interventions: Drug: Propofol; Drug: Fentanyl
- Dexmedetomidine (Active Comparator): Dexmedetomidine will be administered for sedation
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — Propofol will be administered for sedation in mechanically ventilated patients with sepsis.
  Other Names: Diprivan
  Arms: Propofol
Drug: Dexmedetomidine — Dexmedetomidine will be administered for sedation in mechanically ventilated patients with sepsis.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Fentanyl — Fentanyl will be administered for analgesia in mechanically ventilated patients with sepsis. The use of Fentanyl is not an intervention "of interest".

SUMMARY:
Patients with infections in their blood often become very sick. These patients are usually put in an intensive care unit for careful observation and treatment. These patients may develop a low blood pressure, lung failure, and kidney failure. When these problems develop, care becomes quite complicated. Patients with lung failure often need help with a breathing machine to make certain that the breathing is adequate. The machine helps keep the oxygen level high enough for healthy tissues. When patients are placed on the machine for breathing they require a tube to be placed into lungs. This can be quite uncomfortable. These patients need sedation to help them tolerate the uncomfortable breathing tube and other parts of their routine necessary care. This study will compare two drugs (dexmedetomidine and propofol) which are frequently used for sedation in intensive care patients. Clinical studies suggest that these drugs are both effective and safe. The main question is whether or not one of the drugs is better in a patient with a blood infection. This study will try to determine that. Our main goal is to see whether or not patients on one particular drug come off the breathing machine faster than patients on the other drug. These drugs are not experimental drugs and are approved by the Food and Drug Administration. There is no placebo drug being used in this study. All patients in this study will receive the best possible care based on their medical condition.

DETAILED DESCRIPTION:
Patients admitted to the MICU with acute respiratory care and possible sepsis will be evaluated and managed by the internal medicine MICU team. This team includes faculty members, pulmonary fellows, and internal medicine residents. These physicians will make all the decisions regarding the initial management of the patient. The admitting team will be approached by the study investigators to solicit their support for the recruitment of the patient into the study. During some periods of time the study investigators will be directly involved in the patient care.

The general approach to managing patients with sepsis includes blood cultures, serum lactate levels, and empiric antibiotics. Other cultures from the respiratory tract, urinary tract, and other sites are also obtained as indicated. Empiric antibiotic choices will be based on the most likely source of infection. Patient will receive fluid administration and vasopressors to maintain mean arterial pressure blood pressures greater than or equal to 60 mmHg.

Mechanical ventilation support will follow ARDS network guidelines. In general patients will be on an assist-control mode, a low tidal volume (6 mm/kg ideal body weight), and a FiO2 adequate to maintain O2 saturations greater than equal to 90%. PEEP levels will be based on the FiO2 using ARDS network recommendations. The ventilator management goal is to have the lowest possible plateau pressure and lowest FiO2 possible to maintain adequate ventilation and oxygenation.

Fentanyl will be routinely ordered for analgesia. Per current UMC policy, initial fentanyl boluses will be given at 50mcg IV every 2 hours as needed to keep pain level less than 4/10. At the discretion of the provider, a fentanyl drip may be administered if intermittent fentanyl does not achieve adequate analgesia. If a fentanyl drip is initiated, the drip will have a range of 25-200 mcg/hour to achieve a pain level of less than 4/10. If an allergy to fentanyl is documented, the patient will be excluded from the study.

Once a mechanically ventilated patient with sepsis is selected for enrollment, the patient will be randomized (via a computer-generated randomization program) to one of two sedation arms: 1) propofol, or 2) dexmedetomidine.

Per current UMC policy, propofol will be initiated at 5 mcg/kg/minute (0.3mg/kg/hour) and titrated every 5 minutes by 5mcg/kg/minute to RASS (Richmond Agitation and Sedation Scale) goal -1 to +1. The maximum dose of propofol will be 80 mcg/kg/minute.

Dexmedetomidine will be initiated at 0.2 mcg/kg/hour and will be titrated every 5 minutes by 0.1mcg/kg/hour to a maximum dose of 1.4 mcg/kg/hour to a RASS goal of -1 to +1. Although dexmedetomidine has only been approved in the United States for short-term sedation of ICU patients (< 24 hrs) at a maximal dose of 0.7 μg/kg/hr (up to 1.0 μg/kg/h for procedural sedation), several studies demonstrate the safety and efficacy of dexmedetomidine infusions administered for greater than 24 hrs (up to 28 days) and at higher doses (up to 1.5 μg/kg/hr).

Daily sedation stops will be performed in both study arms per MICU weaning policy. Patients will be allowed to return to a RASS of 0 to +1, and the physician will be alerted for assessment. If the physician determines sedation needs to be re-started, it will be at 50% of the dose prior to the sedation stop. This dose will then be titrated to a RASS goal of -1 to +1.

Patients with inadequate sedation scores on their assigned drug will receive supplemental sedation with midazolam or lorazepam using IV boluses as needed based on nursing and physician assessment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-89 years old
* with the diagnosis of sepsis (as specified below) within the previous 24 hours
* who require mechanical ventilation, and
* provide informed consent either personally or by an authorized representative.

Exclusion Criteria:

* Patients with documented allergies to propofol, dexmedetomidine, fentanyl, eggs or egg products, or soy or soy products.
* A heart rate less than 50 beats/minute or grade 2 or 3 AV heart block
* Mean arterial pressure less than 55 mmHg despite appropriate fluid resuscitation and vasopressor support.
* Current triglyceride level > 400 mg/dl

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Nugent, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- University Medical Center, Lubbock, Texas, United States

REFERENCES:
- [Background] Carson SS, Kress JP, Rodgers JE, Vinayak A, Campbell-Bright S, Levitt J, Bourdet S, Ivanova A, Henderson AG, Pohlman A, Chang L, Rich PB, Hall J. A randomized trial of intermittent lorazepam versus propofol with daily interruption in mechanically ventilated patients. Crit Care Med. 2006 May;34(5):1326-32. doi: 10.1097/01.CCM.0000215513.63207.7F. PMID 16540958
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Pandharipande PP, Sanders RD, Girard TD, McGrane S, Thompson JL, Shintani AK, Herr DL, Maze M, Ely EW; MENDS investigators. Effect of dexmedetomidine versus lorazepam on outcome in patients with sepsis: an a priori-designed analysis of the MENDS randomized controlled trial. Crit Care. 2010;14(2):R38. doi: 10.1186/cc8916. Epub 2010 Mar 16. PMID 20233428
- [Background] Jakob SM, Ruokonen E, Grounds RM, Sarapohja T, Garratt C, Pocock SJ, Bratty JR, Takala J; Dexmedetomidine for Long-Term Sedation Investigators. Dexmedetomidine vs midazolam or propofol for sedation during prolonged mechanical ventilation: two randomized controlled trials. JAMA. 2012 Mar 21;307(11):1151-60. doi: 10.1001/jama.2012.304. PMID 22436955
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Result] Sigler MB, Islam EA, Nugent K. Comparison of dexmedetomidine and propofol in mechanically ventilated patients with sepsis: a pilot study. The Southwest Respiratory and Critical Care Chronicles 2018;6(22):10-15.

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol: Propofol will be administered for sedation.
  Propofol: Propofol will be administered for sedation in mechanically ventilated patients with sepsis using a titration based on level of agitation.
  Fentanyl: Fentanyl will be administered for analgesia in mechanically ventilated patients with sepsis. The use of Fentanyl is not an intervention "of interest".
- Dexmedetomidine: Dexmedetomidine will be administered for sedation
  Dexmedetomidine: Dexmedetomidine will be administered for sedation in mechanically ventilated patients with sepsis using a titration based on level of agitation.
  Fentanyl: Fentanyl will be administered for analgesia in mechanically ventilated patients with sepsis. The use of Fentanyl is not an intervention "of interest".
Period: Overall Study
Arm/Group | Propofol | Dexmedetomidine
Started (Duration of mechanical ventilation) | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Dexmedetomidine | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (15.4) | 62.5 (9.6) | 60.75 (NA) — The person who managed this study has left the school and the raw data are not available.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 9 | 13 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.1 (6.5) | 29.7 (8.2) | 29.9 (NA) — The person who managed this study has left the school and the raw data are not available

OUTCOME MEASURES:

1. Primary Outcome: Duration of Mechanical Ventilation
Description: Number of days patient requires mechanical ventilation
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 19 | 17
days | 5 [3 to 13] | 3 [2.75 to 5.75]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Equivalence — Outcome comparison used the Mann Whitney U test; p = 0.107, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Duration of MICU Stay
Description: Number of days patient stays in the MICU
Time Frame: Up to 28 Days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 19 | 17
days | 6 [4 to 14] | 5 [3 to 8]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Equivalence — Outcomes were compared using a Mann Whitney U test; p = 0.260, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Duration of Vasopressor Support
Description: Number of days the patient requires intravenous vasopressors
Time Frame: Up to 28 Days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 19 | 17
days | 0 [0 to 3.3] | 2 [0 to 3]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Equivalence — Outcomes were compared using a Mann Whitney U test; p = 0.376, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mortality
Description: Number of patients who die within 28 days after randomization
Time Frame: Up to 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 19 | 17
Participants | 8 | 9
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Equivalence — Outcomes were compared using a Chi square test; p = 0.739, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 28 days
Arm/Group | Propofol | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 8/19 | 9/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes